CLINICAL TRIAL: NCT05259982
Title: Vital Root-resective Therapy in Furcation-involved Maxillary Molars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Santiago de Compostela (Other)
Responsible Party: Principal Investigator, José Dopico, Clinical Lecturer, University of Santiago de Compostela
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Furca_2
Record Dates: First submitted 2022-02-06; First posted 2022-03-02 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Periodontitis; Furcation Defects
Keywords: Periodontitis; Furcation
MeSH Terms: conditions — Periodontitis; Furcation Defects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vital root resection (Experimental): Root resective surgery aiming to preserve pulp vitality
  Interventions: Procedure: Vital root resection

INTERVENTIONS:
Procedure: Vital root resection — Vital resection of root with attachment loss exceeding 2/3 of the root with the use of calcium silicate cement in the pulpal wound

SUMMARY:
The primary aim of this study is to evaluate 1-year survival of maxillary molars with subclass C vertical furcation involvement after vital root resective therapy

DETAILED DESCRIPTION:
Schedule of Treatment for each visit:

Visit 1 - Baseline (day 0)

* Informed Consent, medical/dental history and demographics
* Record concomitant medications
* Periodontal assessment with recording of full mouth PPD, gingival recession, bleeding on probing (BOP), tooth mobility and furcation involvement
* Long cone periapical radiographs with paralleling technique (if radiograph taken in previous 3 months is not available)
* CBCT examination
* Photographs
* Oral hygiene instructions
* Sensitivity tests

Visit 2 - Treatment (intervention) visit

* Medical/dental history update and record adverse events and/or concomitant medications
* Root-resective surgery
* Post-treatment regime will be outlined according to protocol

Visit 3 - 1 Week Post-Intervention and Further Treatment

* Update medical/dental history and record adverse events and/or concomitant medications
* Clinical photos
* Post-treatment regime will be outlined according to protocol

Visit 4 - 1-Month Post-Intervention

* Update medical/dental history and record adverse events and/or concomitant medications
* Full mouth plaque score (FMPS) recording (6 sites per tooth)
* Oral hygiene reinforcement, full mouth supra-gingival debridement to remove new accumulations of plaque or calcified deposits and supra-gingival polishing
* Clinical photos
* Sensitivity tests

Visit 5 - 3 Months Post-Intervention

* Update medical/dental history and record adverse events and/or concomitant medications
* FMPS recording
* Oral hygiene reinforcement, full mouth supra-gingival debridement to remove new accumulations of plaque or calcified deposits and supra-gingival polishing
* Periodontal assessment consisting of recording of full mouth (6 sites per tooth) PPD, recession, BOP, mobility (tooth level) and furcation involvement (for each multirooted tooth)
* Clinical photos
* Sensitivity tests

Visit 6 - 6 Months Post Intervention

* Update medical/dental history and record adverse events and/or concomitant medications
* Clinical photos
* FMPS recording
* Periodontal assessment consisting of recording of full mouth PPD, recession, BOP, tooth mobility and furcation involvement
* Oral hygiene reinforcement, full mouth supra- and sub-gingival debridement to remove new accumulations of plaque or calcified deposits and supra-gingival polishing
* Sensitivity tests

Visit 7 - 9 Months Post Intervention

* Update medical/dental history and record adverse events and/or concomitant medications
* Clinical photos
* FMPS recording
* Periodontal assessment consisting of recording of full mouth PPD, recession, BOP, tooth mobility and furcation involvement
* Oral hygiene reinforcement, full mouth supra- and sub-gingival debridement to remove new accumulations of plaque or calcified deposits and supra-gingival polishing
* Sensitivity tests

Visit 8 - 12 Months Post Intervention

* Update medical/dental history and record adverse events and/or concomitant medications
* Clinical photos
* FMPS recording
* Periodontal assessment consisting of recording of full mouth PPD, recession, BOP, tooth mobility and furcation involvement
* Oral hygiene reinforcement, full mouth supra- and sub-gingival debridement to remove new accumulations of plaque or calcified deposits and supra-gingival polishing
* Sensitivity tests

Description of study procedures:

Clinical periodontal examination:

Dichotomous (no/yes) full mouth plaque scores (FMPS) will be recorded, identifying tooth surfaces revealing the visual presence of plaque following the use of plaque-disclosing tablets. Periodontal measurements will be taken by the calibrated examiner at six sites per tooth using a manual University of North Carolina (UNC-15) periodontal probe. The following periodontal measurements will be taken full mouth at 6 sites per tooth: probing pocket depth (PPD), recession of the gingival margin from the cemento-enamel junction (CEJ), dichotomous (no/yes) bleeding on probing (BoP). Recession will be recorded as a negative number if the gingival margin is above CEJ; and as a positive number (incl. 0) if margin is on (0) or below CEJ (>0). Further, tooth mobility (no/yes and degree 1, 2 or 3), horizontal furcation involvement using a Nabers probe (no/yes and degree 1, 2 or 3) and finally vertical furcation involvement (no/yes and class A, B or C) measured with a UNC-15 probe will be recorded. Clinical attachment levels (CAL) will be calculated as PPD + recession. This is part of standard care.

Sensitivity testing:

Cold stimulus (Endo-Frost; Roeko GmbH & Co - Coltène-Whaledent, Switzerland) will be applied on a sprayed cotton pellet to the cervical third of the buccal and palatal surfaces of isolated teeth after gentle air-drying and for up to 10 seconds per tooth. A negative response will be recorded when the subject fails to indicate a response on two consecutive occasions on each surface.

Electric testing will be carried out following manufacturer instructions by placing the toothpaste-impregnated probe tip to the occlusal third of the tooth. A plastic interproximal matrix band will be used between teeth to prevent current conduction to the adjacent teeth. A negative response will be recorded when the tester reaches its maximum level on two consecutive occasions.

Root-resective surgery:

Following rinsing with chlorhexidine digluconate 0.12% mouthwash (Perio-Aid; Dentaid, Spain) and administration of local anaesthetic (Xilonibsa 20 mg/ml + 0,0125 mg/ml; Inibsa SA), intrasulcular and/or submarginal incisions will be performed as judged by the clinician. Releasing incisions may be performed if necessary. Full-thickness flaps will be elevated to access the furcation area. Granulation tissue will be eliminated with the aid of curettes (Hu-Friedy Manufacturing Co LLC), and root surface debridement will be performed with ultrasonic devices (EMS, Switzerland) with specific thin and delicate inserts and/or curettes. The root scheduled for resection will be separated from the root using high-speed rotary instruments. Once complete root separation is verified, it will be carefully elevated from the socket. Additional cuts in the separated root may be performed as necessary in order to minimise trauma to the socket and the tooth. Following root resection, the tooth will be isolated with rubber dam and a light-cured resin barrier (Opaldam, Ultradent Products) to avoid contamination of the pulpal wound. A 3-mm amputation of the pulp will be carried out with sterile round diamond burs under water cooling, to allow space for both pulp capping and restorative material. Pressure will be applied on the exposed pulp for up to 5 minutes with a sterile cotton pellet soaked in 2.5% NaOCl to achieve hemostasis. The exposure cavity will be filled with Biodentine (Septodont, Saint Maur des Fossés, France) following manufacturer's instructions on material manipulation and placement. After initial setting of the capping material (12 minutes from mixing), a rubber dam will be placed in order to isolate the resection site and avoid moisture, and 1 mm of Biodentine will be removed with a sterile tungsten carbide bur at low speed (5000-10000 rpm) under copious irrigation. A self-etching dentine adhesive (Clearfil SE Bond; Kuraray, Osaka, Japan) will be applied to the cavity and subsequently restored with a light-cured resin composite (Clearfil AP-X; Kuraray, Osaka Japan). Finishing and polishing of the restoration will be accomplished with a very fine diamond bur. Careful recontouring of the resection area will be performed in order to avoid ledges or plaque-retentive anatomy. Bone resection will be performed with rotary and manual instruments as judged by the clinician. Flaps will be will be repositioned and sutured with 5/0 and 6/0 monofilament sutures (Seralene; Serag-Wiessner GmbH & Co. KG). Gentle pressure will be applied with a moist gauze until haemostasis is achieved.

Follow-up Procedures:

All sites in the mouth of participants will receive the required periodontal treatment by a trained therapist (periodontist/dentist/hygienist) throughout the duration of the study, as judged by the examining clinician. This is likely to involve supportive periodontal therapy (including supra- and sub-gingival debridement, polishing, oral hygiene re-enforcements and motivation) but may also involve more advanced periodontal treatment including surgical options. If any participant-related acute medical or dental problems arise, these will be managed in the appropriate manner in line with routine clinical practice. Where appropriate, if care is required in relation to one of the study treatment procedures, participants will be seen at the study site. In other cases, following an assessment of the most appropriate treatment required, participants will be appropriately directed to their medical or dental general practitioner.

At the study completion phase the patient may be further allocated for treatment if it is deemed necessary. If no such treatment is required then the patient will be enrolled in a supportive periodontal therapy program.

'Rescue' therapy: In case of continued CAL >2mm at 2 consecutive appointments, an extra session of sub-gingival debridement under local anaesthesia or an access flap operation will be planned for the study site, as judged by the examining clinician. In case of development of endodontic pathology: consider endodontic therapy (if indicated) or otherwise extraction (if combined with mobility > I). In the case of a development of root fracture or in cases of excessive mobility or patient discomfort, extraction will be considered and discussed with the patient. Any further treatment carried out on the molar with FI will be recorded and analysed. If any extraction is carried out, the reason for extraction will be documented in the case-report forms.

In case endodontic pathology developed, the patient will be provided endodontic treatment.

Radiographic Assessments:

The selected study defect will be detected based on radiographs often taken at the new patient consultation or provided by referring dentists. A long-cone periapical radiograph of selected study sites will be taken by one of the study investigators at baseline, 6 and 12-month follow-up visits. Additional radiographs may be taken when considered clinically necessary by the treating clinician.

These radiographs are considered standard of care as they will be important for treatment planning purposes and for assessing the treatment response. They will also help decide whether or not the teeth are still maintainable post-treatment.

A preoperative limited-volume CBCT will be taken in order to assess root morphology and presence of periapical pathology. A follow-up CBCT scan will be taken at 12 months in order to assess the presence of periapical pathology and intra-pulpal calcifications in reaction to the treatment.

ELIGIBILITY:
Inclusion Criteria

* Minimum of 12 teeth present
* Diagnosis of Severe Periodontitis stage III or IV (Tonetti et al., 2018)
* At least one maxillary molar with: i) degree II-III horizontal furcation involvement (Eickholz and Walter, 2018), ii) class C vertical furcation involvement (bone loss up to the apical third of root cones) (Tarnow and Fletcher, 1984, Tonetti et al., 2017), iii) residual probing pocket depths > 5 mm, iv) maximum mobility degree I (Hamp et al., 1975) and v) not already accessible for self-performed oral hygiene
* Received a course of non-surgical periodontal therapy within the past six months
* Positive response to electric and cold testing

Exclusion Criteria

Patient:

* Full mouth plaque score > 30%
* A course of antibiotics within the past 3 months
* Pregnant/lactating women
* Relevant medical history as evaluated by the examining clinician which may have the potential to affect periodontal surgical treatment (such as disease affecting clotting ability)
* Individuals on long-standing (2 or above years) supportive periodontal therapy (SPT) management plans

Molar affected by FI:

* Ongoing endodontic pathology affecting the furcation-involved molar, as judged by the examining clinician
* Teeth associated with signs or symptoms indicative of pulpal or periapical pathology
* Evidence of coronal cracks upon root resection
* Previous periodontal surgical treatment to the furcation-affected molar within the previous 5 years
* Endodontically treated tooth
* Restorations affecting more than 2 walls or 1 cusp
* Molar tooth acting as a bridge abutment
* Planned for extraction (for strategic/restorative reasons)
* Root trunk exceeding ½ of the total root length
* Fused roots
* Remaining furcation not accessible for self-performed oral hygiene
* The presence of occlusal dysfunction as assessed by the examining clinician
* Sinus floor anatomy limiting possible osseous resective surgery
* Tooth mobility causing discomfort to the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-03-04 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Tooth survival | 1 year
  Tooth present or absent after treatment (yes/no)

SECONDARY OUTCOMES:
Probing pocket depth | 1 year
  Distance from gingival margin to deepest point of the pocket
Clinical attachment levels | 1 year
  Distance from CEJ to deepest point of the pocket
Radiographic bone levels | 1 year
  Periapical radiographs and/or CBCT
Pulpal response to sensitivity tests | 1 year
  Positive or negative response to electric and cold pulp tests (yes/no).
  Cold stimulus (Endo-Frost; Roeko GmbH & Co - Coltène-Whaledent, Switzerland) will be applied on a sprayed cotton pellet to the cervical third of the buccal and palatal surfaces of isolated teeth after gentle air-drying and for up to 10 seconds per tooth. A negative response will be recorded when the subject fails to indicate a response on two consecutive occasions on each surface.
  Electric testing will be carried out following manufacturer instructions by placing the toothpaste-impregnated probe tip to the occlusal third of the tooth. A plastic interproximal matrix band will be used between teeth to prevent current conduction to the adjacent teeth. A negative response will be recorded when the tester reaches its maximum level on two consecutive occasions.
Clinical signs or symptoms indicative of periapical pathology | 1 year
  Periapical radiolucencies, sinus tract, swelling, tenderness to percussion, coronal discolouration, pain on biting, cold and heat lingering sensitivity, persistent or spontaneous dull throbbing pain
Formation of calicified tissue in the pulp exposure | 1 year
  Presence or absence of radio-opaque area over pulp exposure assessed on CBCT (yes/no)
Tooth mobility | 1 year
  Yes/no
Further treatment needed | 1 year
  e.g. repeated instrumentation, prosthetic intervention, etc

CONTACTS AND LOCATIONS:
Overall Officials: José L Dopico García, Dr, Principal Investigator — Universidad de Santiago de Compostela
Locations (1):
- Facultad de Odontologia, Santiago de Compostela, Coruña, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Albandar JM. A 6-year study on the pattern of periodontal disease progression. J Clin Periodontol. 1990 Aug;17(7 Pt 1):467-71. doi: 10.1111/j.1600-051x.1990.tb02346.x. PMID 2403413
- [Background] Brizuela C, Ormeno A, Cabrera C, Cabezas R, Silva CI, Ramirez V, Mercade M. Direct Pulp Capping with Calcium Hydroxide, Mineral Trioxide Aggregate, and Biodentine in Permanent Young Teeth with Caries: A Randomized Clinical Trial. J Endod. 2017 Nov;43(11):1776-1780. doi: 10.1016/j.joen.2017.06.031. Epub 2017 Sep 14. PMID 28917577
- [Background] Carnevale G, Di Febo G, Tonelli MP, Marin C, Fuzzi M. A retrospective analysis of the periodontal-prosthetic treatment of molars with interradicular lesions. Int J Periodontics Restorative Dent. 1991;11(3):189-205. No abstract available. PMID 1802876
- [Background] Chen MX, Zhong YJ, Dong QQ, Wong HM, Wen YF. Global, regional, and national burden of severe periodontitis, 1990-2019: An analysis of the Global Burden of Disease Study 2019. J Clin Periodontol. 2021 Sep;48(9):1165-1188. doi: 10.1111/jcpe.13506. Epub 2021 Jul 7. PMID 34101223
- [Background] Dommisch H, Walter C, Dannewitz B, Eickholz P. Resective surgery for the treatment of furcation involvement: A systematic review. J Clin Periodontol. 2020 Jul;47 Suppl 22:375-391. doi: 10.1111/jcpe.13241. PMID 31912534
- [Background] Dopico J, Nibali L, Donos N. Disease progression in aggressive periodontitis patients. A Retrospective Study. J Clin Periodontol. 2016 Jun;43(6):531-7. doi: 10.1111/jcpe.12533. Epub 2016 May 2. PMID 26878438
- [Background] Filipowicz F, Umstott P, England M. Vital root resection in maxillary molar teeth: a longitudinal study. J Endod. 1984 Jun;10(6):264-8. doi: 10.1016/S0099-2399(84)80060-6. No abstract available. PMID 6590730
- [Background] Graetz C, Schutzhold S, Plaumann A, Kahl M, Springer C, Salzer S, Holtfreter B, Kocher T, Dorfer CE, Schwendicke F. Prognostic factors for the loss of molars--an 18-years retrospective cohort study. J Clin Periodontol. 2015 Oct;42(10):943-50. doi: 10.1111/jcpe.12460. Epub 2015 Oct 26. PMID 26399690
- [Background] Guerrero A, Griffiths GS, Nibali L, Suvan J, Moles DR, Laurell L, Tonetti MS. Adjunctive benefits of systemic amoxicillin and metronidazole in non-surgical treatment of generalized aggressive periodontitis: a randomized placebo-controlled clinical trial. J Clin Periodontol. 2005 Oct;32(10):1096-107. doi: 10.1111/j.1600-051X.2005.00814.x. PMID 16174275
- [Background] Hamp SE, Nyman S, Lindhe J. Periodontal treatment of multirooted teeth. Results after 5 years. J Clin Periodontol. 1975 Aug;2(3):126-35. doi: 10.1111/j.1600-051x.1975.tb01734.x. PMID 1058213
- [Background] Hashem D, Mannocci F, Patel S, Manoharan A, Brown JE, Watson TF, Banerjee A. Clinical and radiographic assessment of the efficacy of calcium silicate indirect pulp capping: a randomized controlled clinical trial. J Dent Res. 2015 Apr;94(4):562-8. doi: 10.1177/0022034515571415. Epub 2015 Feb 20. PMID 25710953
- [Background] Haskell EW. Vital root resection on maxillary multi-rooted teeth. J South Calif Dent Assoc. 1966 Nov;34(11):509-12. No abstract available. PMID 5224492
- [Background] Haskell EW. Vital root resection. Oral Surg Oral Med Oral Pathol. 1969 Feb;27(2):266-74. doi: 10.1016/0030-4220(69)90182-0. No abstract available. PMID 5249524
- [Background] Hegde S, Sowmya B, Mathew S, Bhandi SH, Nagaraja S, Dinesh K. Clinical evaluation of mineral trioxide aggregate and biodentine as direct pulp capping agents in carious teeth. J Conserv Dent. 2017 Mar-Apr;20(2):91-95. doi: 10.4103/0972-0707.212243. PMID 28855754
- [Background] Huynh-Ba G, Kuonen P, Hofer D, Schmid J, Lang NP, Salvi GE. The effect of periodontal therapy on the survival rate and incidence of complications of multirooted teeth with furcation involvement after an observation period of at least 5 years: a systematic review. J Clin Periodontol. 2009 Feb;36(2):164-76. doi: 10.1111/j.1600-051X.2008.01358.x. PMID 19207893
- [Background] Jepsen K, Dommisch E, Jepsen S, Dommisch H. Vital root resection in severely furcation-involved maxillary molars: Outcomes after up to 7 years. J Clin Periodontol. 2020 Aug;47(8):970-979. doi: 10.1111/jcpe.13306. Epub 2020 Jun 8. PMID 32412133
- [Background] Kassebaum NJ, Bernabe E, Dahiya M, Bhandari B, Murray CJ, Marcenes W. Global Burden of Severe Tooth Loss: A Systematic Review and Meta-analysis. J Dent Res. 2014 Jul;93(7 Suppl):20S-28S. doi: 10.1177/0022034514537828. PMID 24947899
- [Background] Linu S, Lekshmi MS, Varunkumar VS, Sam Joseph VG. Treatment Outcome Following Direct Pulp Capping Using Bioceramic Materials in Mature Permanent Teeth with Carious Exposure: A Pilot Retrospective Study. J Endod. 2017 Oct;43(10):1635-1639. doi: 10.1016/j.joen.2017.06.017. Epub 2017 Aug 12. PMID 28807371
- [Background] Low KM, Dula K, Burgin W, von Arx T. Comparison of periapical radiography and limited cone-beam tomography in posterior maxillary teeth referred for apical surgery. J Endod. 2008 May;34(5):557-62. doi: 10.1016/j.joen.2008.02.022. PMID 18436034
- [Background] Nibali L, Krajewski A, Donos N, Volzke H, Pink C, Kocher T, Holtfreter B. The effect of furcation involvement on tooth loss in a population without regular periodontal therapy. J Clin Periodontol. 2017 Aug;44(8):813-821. doi: 10.1111/jcpe.12756. Epub 2017 Jul 12. PMID 28699678
- [Background] Nibali L, Yeh YC, Pometti D, Tu YK. Long-term stability of intrabony defects treated with minimally invasive non-surgical therapy. J Clin Periodontol. 2018 Dec;45(12):1458-1464. doi: 10.1111/jcpe.13021. Epub 2018 Nov 5. PMID 30307641
- [Background] Nibali L, Zavattini A, Nagata K, Di Iorio A, Lin GH, Needleman I, Donos N. Tooth loss in molars with and without furcation involvement - a systematic review and meta-analysis. J Clin Periodontol. 2016 Feb;43(2):156-66. doi: 10.1111/jcpe.12497. Epub 2016 Feb 12. PMID 26932323
- [Background] Nowicka A, Lipski M, Parafiniuk M, Sporniak-Tutak K, Lichota D, Kosierkiewicz A, Kaczmarek W, Buczkowska-Radlinska J. Response of human dental pulp capped with biodentine and mineral trioxide aggregate. J Endod. 2013 Jun;39(6):743-7. doi: 10.1016/j.joen.2013.01.005. Epub 2013 Apr 10. PMID 23683272
- [Background] Papapanou PN, Sanz M, Buduneli N, Dietrich T, Feres M, Fine DH, Flemmig TF, Garcia R, Giannobile WV, Graziani F, Greenwell H, Herrera D, Kao RT, Kebschull M, Kinane DF, Kirkwood KL, Kocher T, Kornman KS, Kumar PS, Loos BG, Machtei E, Meng H, Mombelli A, Needleman I, Offenbacher S, Seymour GJ, Teles R, Tonetti MS. Periodontitis: Consensus report of workgroup 2 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Clin Periodontol. 2018 Jun;45 Suppl 20:S162-S170. doi: 10.1111/jcpe.12946. PMID 29926490
- [Background] Papapanou PN, Tonetti MS. Diagnosis and epidemiology of periodontal osseous lesions. Periodontol 2000. 2000 Feb;22:8-21. doi: 10.1034/j.1600-0757.2000.2220102.x. No abstract available. PMID 11276518
- [Background] Patel S, Wilson R, Dawood A, Foschi F, Mannocci F. The detection of periapical pathosis using digital periapical radiography and cone beam computed tomography - part 2: a 1-year post-treatment follow-up. Int Endod J. 2012 Aug;45(8):711-23. doi: 10.1111/j.1365-2591.2012.02076.x. PMID 22775142
- [Background] Pretzl B, Eickholz P, Saure D, Pfefferle T, Zeidler A, Dannewitz B. Endodontic status and retention of molars in periodontally treated patients: results after 10 or more years of supportive periodontal therapy. J Clin Periodontol. 2016 Dec;43(12):1116-1123. doi: 10.1111/jcpe.12621. Epub 2016 Oct 17. PMID 27570936
- [Background] Smukler H, Tagger M. Vital root amputation. A clinical and histological study. J Periodontol. 1976 Jun;47(6):324-30. doi: 10.1902/jop.1976.47.6.324. PMID 1064719
- [Background] Svardstrom G, Wennstrom JL. Prevalence of furcation involvements in patients referred for periodontal treatment. J Clin Periodontol. 1996 Dec;23(12):1093-9. doi: 10.1111/j.1600-051x.1996.tb01809.x. PMID 8997653
- [Background] Tahmooressi K, Jonasson P, Heijl L. Vital root resection with MTA: a pilot study. Swed Dent J. 2016;40(1):43-51. PMID 27464381
- [Background] Tarnow D, Fletcher P. Classification of the vertical component of furcation involvement. J Periodontol. 1984 May;55(5):283-4. doi: 10.1902/jop.1984.55.5.283. PMID 6588186
- [Background] Tonetti MS, Christiansen AL, Cortellini P. Vertical subclassification predicts survival of molars with class II furcation involvement during supportive periodontal care. J Clin Periodontol. 2017 Nov;44(11):1140-1144. doi: 10.1111/jcpe.12789. Epub 2017 Sep 22. PMID 28771794
- [Background] Tonetti MS, Claffey N; European Workshop in Periodontology group C. Advances in the progression of periodontitis and proposal of definitions of a periodontitis case and disease progression for use in risk factor research. Group C consensus report of the 5th European Workshop in Periodontology. J Clin Periodontol. 2005;32 Suppl 6:210-3. doi: 10.1111/j.1600-051X.2005.00822.x. No abstract available. PMID 16128839
- [Background] Tonetti MS, Greenwell H, Kornman KS. Staging and grading of periodontitis: Framework and proposal of a new classification and case definition. J Clin Periodontol. 2018 Jun;45 Suppl 20:S149-S161. doi: 10.1111/jcpe.12945. PMID 29926495
- [Background] White DA, Tsakos G, Pitts NB, Fuller E, Douglas GV, Murray JJ, Steele JG. Adult Dental Health Survey 2009: common oral health conditions and their impact on the population. Br Dent J. 2012 Dec;213(11):567-72. doi: 10.1038/sj.bdj.2012.1088. PMID 23222333